CLINICAL TRIAL: NCT06012773
Title: Investigation of the Relationship Between Neck Posture and Stiffness of Head and Neck Muscles, Pain and Proprioception in Desk Workers
Brief Title: Relationship Between Neck Posture and Stiffness of Head and Neck Muscles, Pain and Proprioception in Desk Workers
Status: Completed | Type: Observational
Sponsor: Pınar Kuyulu (Other)
Responsible Party: Sponsor-Investigator, Pınar Kuyulu, Director, Sanko University
Organization: Sanko University (Other)
Other Study IDs: 2021/01
Record Dates: First submitted 2023-08-22; First posted 2023-08-25 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Work-Related Condition; Musculoskeletal Health
Keywords: proprioception; pain; neck posture; neck muscle stiffness; desk worker
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In our study, posture in desk workers; it aims to evaluate the relationship between cervical range of motion, proprioception, muscle stiffness, posture and pain.

DETAILED DESCRIPTION:
One hundred twelve participants were included in the study.

Cervical range of motion and cervical proprioception were evaluated with a cervical range of motion (CROM) goniometer device, and muscle stiffness was evaluated with myotonometer device. Pain was evaluated with visual analog scale, and Migraine disability assessment scale (MIDAS) and Neck disability index.

Posture was evaluated with Posture Screen mobile application.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer individuals aged 18-65
* Individuals using a computer in a sitting position at a desk

Exclusion Criteria:

* Individuals who have had serious traumatic injuries to the head, neck and shoulder area
* Individuals who have undergone any surgery on the head, neck and shoulder region
* Individuals with any anomaly in the head, neck and shoulder region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Office workers
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
neck proprioception | 20 months
  Cervical range of motion and cervical proprioception were evaluated with a cervical range of motion (CROM) goniometer device.
Neck region muscle stiffness | 20 months
  stiffness of head and neck muscles stiffness was evaluated with myotonometer device.
Neck posture | 20 months
  Posture was evaluated with Posture Screen mobile application.
Cervical range of motion | 20 months
  Cervical range of motion and cervical proprioception were evaluated with a cervical range of motion (CROM) goniometer device.

SECONDARY OUTCOMES:
Head and neck pain | 20 months
  Pain was evaluated with visual analog scale, and Migraine disability assessment scale (MIDAS) and Neck disability index.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Uzun, PhD(c), Principal Investigator — Sanko University
Locations (1):
- SANKO University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No